CLINICAL TRIAL: NCT02127541
Title: New Imaging Procedure for the Localisation of Insulinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other); Desirée and Niels Yde's Foundation, Zürich, Switzerland (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: EKBB 163/12
Record Dates: First submitted 2014-02-10; First posted 2014-04-30 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Endogenous Hyperinsulinaemic Hypoglycaemia
Keywords: Localisation of Insulinoma; beta-cell imaging; exendin-4; 68Ga-DOTA-exendin-4 PET/CT; 111In-DOTA-exendin-4 SPECT/CT
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; 68Ga-DOTA-exendin-4

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ga -exendin PET/CT, In- exendin SPECT/CT, MRI (Experimental): This is a cross-over study comparing three imaging methods (68Ga-DOTA-exendin-4 PET/CT, 111In-DOTA-exendin-4 SPECT/CT, MRI) in the same patient.
  Interventions: Other: Ga -exendin PET/CT, In- exendin SPECT/CT, MRI

INTERVENTIONS:
Other: Ga -exendin PET/CT, In- exendin SPECT/CT, MRI — Comparison of different imaging modalities
  Other Names: 68Ga-DOTA-exendin-4; 111In-DOTA-exendin-4; MRI

SUMMARY:
Insulinoma: Insulinoma are rare, small insulin secreting neuroendocrine tumors. The only curative approach is the surgical excision. The preoperative detection remains a challenge. A non-invasive, highly sensitive tool in localizing the insulinomas would be appreciated in the preoperative work-up of these patients. To this aim Glucagon-like peptide-1 receptor (GLP-1R) imaging (Single Photon Emission Computer Tomography co-registered with a CT; SPECT/CT) could be a convenient tool. The possibly more sensitive approach of targeting GLP-1R using Positron emission tomography (PET/CT) methodology has not been investigated in patients so far.

ELIGIBILITY:
Inclusion Criteria:

* Biochemically proven endogenous hyperinsulinaemic hypoglycaemia in the fasting state with neuroglycopenic symptoms or autologous Islet Cell transplantation in the forearm
* Conventional imaging (CT,MRI or EUS) not older than 2 months
* Signed written consent
* Age above 18 years

Exclusion Criteria:

* Kidney failure (creatinine > 140micromol/l)
* Known allergies against Exendin-4 (Byetta or Bydureon)
* Pregnancy
* Breastfeeding
* Medication with Byetta or Bydureon
* Evidence for malignancy (extrapancreatic tumor manifestations)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-01-06; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Measuring Tumour to Background Ratio | 4 years
Measuring the accuracy of the Tumour-Localisation of 68-DOTA-Exendin-4 PET/CT and 111 In-DOTA-exendin-4 SPECT/CT. | 4 years

SECONDARY OUTCOMES:
Accuracy of tumour localisation of standardized MRI in comparison with 68-DOTA-Exendin-4 PET/CT and 111 In-DOTA-exendin-4 SPECT/CT | 4 years
Sensitivity of tumour localisation with 68-DOTA-Exendin-4 PET/CT, 111 In-DOTA-exendin-4 SPECT/CT and standardized MRI in comparison with conventional imaging (CT,MRI and EUS) | 4 years
Evaluation of the side effects of 68Ga-DOTA-exendin-4 and 111In-DOTA-exendin-4 | 4 years
  Through measurement of blood glucose and Quantification of Nausea respectively vomiting by means of the common toxicity criteria score system
Evaluation of the interobserver variability of 68Ga-DOTA-Exendin-4 PET/CT and 111In-DOTA-exendin-4 SPECT/CT | 4 years
Comparison of the angiogenesis markers with the those of breast carcinoma patients | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Damian Wild, MD, PhD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Background] Wild D, Macke H, Christ E, Gloor B, Reubi JC. Glucagon-like peptide 1-receptor scans to localize occult insulinomas. N Engl J Med. 2008 Aug 14;359(7):766-8. doi: 10.1056/NEJMc0802045. No abstract available. PMID 18703486
- [Background] Christ E, Wild D, Forrer F, Brandle M, Sahli R, Clerici T, Gloor B, Martius F, Maecke H, Reubi JC. Glucagon-like peptide-1 receptor imaging for localization of insulinomas. J Clin Endocrinol Metab. 2009 Nov;94(11):4398-405. doi: 10.1210/jc.2009-1082. Epub 2009 Oct 9. PMID 19820010
- [Background] Pattou F, Kerr-Conte J, Wild D. GLP-1-receptor scanning for imaging of human beta cells transplanted in muscle. N Engl J Med. 2010 Sep 23;363(13):1289-90. doi: 10.1056/NEJMc1004547. No abstract available. PMID 20860517
- [Background] Christ E, Wild D, Ederer S, Behe M, Nicolas G, Caplin ME, Brandle M, Clerici T, Fischli S, Stettler C, Ell PJ, Seufert J, Gloor B, Perren A, Reubi JC, Forrer F. Glucagon-like peptide-1 receptor imaging for the localisation of insulinomas: a prospective multicentre imaging study. Lancet Diabetes Endocrinol. 2013 Oct;1(2):115-22. doi: 10.1016/S2213-8587(13)70049-4. Epub 2013 Jul 25. PMID 24622317
- [Derived] Antwi K, Nicolas G, Fani M, Heye T, Pattou F, Grossman A, Chanson P, Reubi JC, Perren A, Gloor B, Vogt DR, Wild D, Christ E. 68Ga-Exendin-4 PET/CT Detects Insulinomas in Patients With Endogenous Hyperinsulinemic Hypoglycemia in MEN-1. J Clin Endocrinol Metab. 2019 Dec 1;104(12):5843-5852. doi: 10.1210/jc.2018-02754. PMID 31298706
- [Derived] Valente LG, Antwi K, Nicolas GP, Wild D, Christ E. Clinical presentation of 54 patients with endogenous hyperinsulinaemic hypoglycaemia: a neurological chameleon (observational study). Swiss Med Wkly. 2018 Nov 18;148:w14682. doi: 10.4414/smw.2018.14682. eCollection 2018 Nov 5. PMID 30449018
- [Derived] Antwi K, Fani M, Heye T, Nicolas G, Rottenburger C, Kaul F, Merkle E, Zech CJ, Boll D, Vogt DR, Gloor B, Christ E, Wild D. Comparison of glucagon-like peptide-1 receptor (GLP-1R) PET/CT, SPECT/CT and 3T MRI for the localisation of occult insulinomas: evaluation of diagnostic accuracy in a prospective crossover imaging study. Eur J Nucl Med Mol Imaging. 2018 Dec;45(13):2318-2327. doi: 10.1007/s00259-018-4101-5. Epub 2018 Jul 28. PMID 30054698